CLINICAL TRIAL: NCT03864796
Title: Detection of Possible Role of CD11a in Pathogenesis of Primary Immune Thrombocytopenia and Effect of Immunosuppressive Therapy on Its Level
Brief Title: Role of CD11a in Pathogenesis of Primary ITP and Effect of Immunosuppressive Therapy on Its Level
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MonaIbraheem Mostafa, clinical research, Assiut University
Other Study IDs: CD11a in ITP
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cases of newly diagnosed ITP: no intervention
- cases of ITP after responding to treatment: no intervention
- healthy subjects: no intervention

SUMMARY:
1. The purpose of this study is to investigate the expression of CD11a on subpopulation of lymphocytes and compared its expression between ITP patients and healthy controls and explores its possible role in the pathogenesis of ITP.
2. this may help in decision to use inhibitors (have been developed to block ICAM-1/LFA-1 interactions,) as a line of treatment for ITP and some of these molecules have reached clinical trials.
3. to study if there is correlation between level of CD11a and severity of bleeding at presentation (estimated by bleeding score defined by British Journal of Haematology 2007 and platelet count)
4. to study effect of immunosuppressive treatment on the level of CD11a by evaluating levels of CD11a after response to treatment.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an autoimmune disease characterized by low platelet counts with or without mucocutaneous bleeding (McMillan 2007).

Like the majority of autoimmune diseases, ITP is an organ-specific disease and abnormalities in the regulation of immune system have been shown to play an important role in the initiation and/or perpetuation of the disease Autoantibodies reacting against platelet glycoproteins can mediate platelet destruction by the monocyte-macrophage system as well as suppress megakaryocyte proliferation and maturation Although auto reactive B lymphocytes secreting antiplatelet antibodies are considered as the main defect, substantial evidence suggests that a generalized dysfunction of auto reactive T cells is the critical immunopathological cause of ITP and the antiplatelet autoantibodies are under the control of T cells and the cytokines they produce Lymphocyte function associated antigen-1 (LFA-1) belonging to the integrin family is composed of the alpha chain CD11a and beta chain CD18 heterologous dimers , and expressed on the surface of T lymphocytes, B lymphocytes, monocytes, macrophages and neutrophils. Its major ligand, intercellular adhesion molecule-1(ICAM-1) , belongs to the immunoglobulin superfamily, distributed on the surface of antigen- presenting cells (APCs) The combination of LFA-1 and ICAM-1 can provide coordinated stimulus signal and promote lymphocyte activation, proliferation and differentiation. In the interaction of T cells with antigen- presenting cells (APCs), LFA-1 and its adaptor ICAM-1 directly participate in the formation of immunological synapse that promotes costimulatory function, leading to increased T cell proliferation and cytotoxicity CD11a is critical for lymphocyte entry into the lymph nodes and normal development of hematopoietic intermediates The disruption of LFA-1 activity strongly affects the stability of immune interface .

The expression of ICAM-1 and LFA-1 is significantly higher on lymphoid cells and vascular endothelial cells in rheumatoid arthritis (RA), indicating that the combination of LFA-1 and ICAM-1 may play an important role in the progression of RA The excessive expression of LFA-1 can induce the formation of auto-reactive T cells, resulting in lupus disease in mice. By using LFA-1 monoclonal antibodies in lupus mice the production of autoantibodies could be reduced, the development of autoimmune reaction stopped, and the symptoms of lupus nephritis alleviated. Therefore, LFA-1 may play an important role in the pathogenesis of systemic lupus erythematosus.

In ITP patients CD11a could facilitate the survival of CD19+ B cells and promote antibody-mediated platelets destruction .Therefore, blocking ICAM-1/LFA-1 interaction can suppress T-cell activation in autoimmune diseases. Many types of inhibitors (i.e. antibodies, peptides, small molecules) have been developed to block ICAM-1/LFA-1 interactions, and some of these molecules have reached clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed primary immune thrombocytopenic patients

Exclusion Criteria:

* We will exclude patients with any other possible cause of thrombocytopenia either immune or non immune as:
* Patients with diabetes
* HCV
* other autoimmune disease (as SLE or RA)
* Chronic Liver or kidney disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people with newely diagnosed primary ITP and healthy control
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
detection of possible role of CD11a in pathogenesis of ITP | 1 year
  assaying of CD11a in patients and healthy individual
detection of effect of immunosuppressive therapy on the level of CD11a in patients of ITP | 1 year
  to study effect of immunosuppressive treatment on the level of CD11a by evaluating levels of CD11a after response to treatment.to detect possible role of CD11a-ICAM1 blocker in treatment of ITP

CONTACTS AND LOCATIONS:
Overall Officials: Howwaida AH Nafady, Prof., Study Director — Assiut University
Locations (1):
- Mona, Asyut, Egypt